CLINICAL TRIAL: NCT02846961
Title: Occurrence of Anti-drug Antibody and Change of Drug Level for 1 Year After CT-P13 Therapy and Their Impact on Clinical Outcomes in Moderate to Severe Inflammatory Bowel Disease (OACIS Study)
Brief Title: Anti CT-P13 Antibody in Moderate to Severe Inflammatory Bowel Disease
Acronym: OACIS
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Other Study IDs: KMU160306
Record Dates: First submitted 2016-07-23; First posted 2016-07-27 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn's Disease
Keywords: inflammatory bowel disease; biosimilar; anti-drug antibody; trough drug concentration
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crohn's disease: Patients with moderate to severe Crohn's disease who need to get a biosimilar CT-P13
- Ulcerative colitis: Patients with moderate to severe ulcerative colitis who need to get a biosimilar CT-P13

SUMMARY:
The purpose of this study is to evaluate the development of anti-drug antibody to biosimilar CT-P13 and to assess the change of drug concentration for 1 year in patients with moderately to severe inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's disease or ulcerative colitis

Exclusion Criteria:

* Tuberculosis infection
* Allergy to CT-P13

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe inflammatory bowel disease who need to receive biosimilar CT-P13
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Development of anti-drug antibody to CT-P13 | one year

SECONDARY OUTCOMES:
Change of drug trough concentration | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Il Park, MD, Study Chair — Sungkyunkwan University
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided